CLINICAL TRIAL: NCT06294353
Title: A Randomized, Multicenter, Treatment-as-usual Controlled Clinical Trial to Evaluate the Safety and Efficacy of Digital Cognitive Behavioral Therapy for Eating Disorder
Brief Title: Study of Efficacy and Safety of WELT-ED for Eating Disorder (WCTP-ED-B-01)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WELT corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCTP-ED-B-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Eating Disorders; Binge Eating; Binge-Eating Disorder
Keywords: Digital Therapeutics; Digital Cognitive Behaviorial Therapy; App Based Intervention
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WELT-ED (CBT based DTx) (Experimental): Participants in this group will receive a shortened version of the standard treatment plus access to the DTx app for 8 weeks.
  The DTx app is designed to provide therapeutic interventions based on CBT principles, aiming to help participants manage and reduce their eating disorder symptoms.
  Participants are expected to engage with the app, completing tasks such as self-monitoring food diaries. The app will collect data on adherence, including diary completion rates and app login frequency.
  Additional Support: Aside from app usage, participants will receive counseling and support therapy during visits at baseline, the 4-week mark, and the 8-week mark.
  They will continue any pre-existing medication for eating disorders.
  Interventions: Device: WELT-ED (CBT based DTx)
- Standard Treatment (Other): Participants will receive the standard treatment protocol for eating disorders, which includes regular counseling and support therapy at all scheduled visits.
  This treatment is comprehensive and follows the conventional approach to managing eating disorders, without the use of the DTx app.
  Participants will continue any pre-existing medication for eating disorders.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Device: WELT-ED (CBT based DTx) — The product delivers Cognitive Behavioral Therapy for Eating Disorders (CBT-ED) through a software interface (iOS and Android), designed to engage patients in a structured and interactive manner. It operates by analyzing patterns in the patient's lifestyle and eating data, identifying problematic behaviors associated with their eating disorder. Based on this analysis, the software sets daily learning objectives aimed at fostering positive cognitive and behavioral habits. By providing tailored guidance and support, the product seeks to assist patients in making sustainable changes, ultimately contributing to the improvement of eating disorder symptoms. This approach combines the principles of CBT-ED with the convenience and accessibility of digital technology, offering a personalized therapeutic experience to support patients in their recovery.
  Arms: WELT-ED (CBT based DTx)
Behavioral: Standard Treatment — In the control group, from screening/baseline (Visit 1) to 8 weeks (Visit 5), counseling and support therapy will be conducted at all visits. Participants can continue taking SSRI medications and other antipsychotic drugs that they were already taking for the treatment of eating disorders during the trial period. However, the intake of any additional antipsychotic drugs, other than those already being taken (including SSRIs), is prohibited during the trial period.
  Arms: Standard Treatment

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of a digital therapeutic device (WELT-ED) based on Cognitive Behavioral Therapy (CBT) for the treatment of eating disorders.

The main questions it aims to answer are:

* Is WELT-ED as effective as standard treatment in reducing the symptoms of eating disorders?
* Is the WELT-ED safe for use in the target population without causing adverse effects?

Participants will:

* Undergo assessments to determine their baseline health status and severity of eating disorder symptoms.
* Use WELT-ED or receive standard treatment as directed for the duration of the study period (8 weeks).
* Participate in assessments to monitor changes in their eating disorder symptoms and any potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 19 and 65 years
* Diagnosed with an eating disorder according to ICD-10.

F50.0 Anorexia nervosa F50.1 Atypical anorexia nervosa F50.2 Bulimia nervosa F50.3 Atypical bulimia nervosa F50.4 Overeating associated with other psychological disturbances F50.5 Vomiting associated with other psychological disturbances F50.8 Other eating disorders F50.9 Eating disorder, unspecified)

* Have a binge eating frequency (as per item 14 of the EDE-Q) of 4 or more times over the past 4 weeks (28 days) at the time of screening.
* Able to use a mobile application (app) on a smartphone without difficulty.
* After receiving and understanding sufficient information about this clinical trial, voluntarily decides to participate and provides written consent.

Exclusion Criteria:

* Previously received Cognitive Behavioral Therapy for the treatment of an eating disorder.
* Have a history of bariatric surgery (e.g., adjustable gastric band, sleeve gastrectomy, biliopancreatic diversion, Roux-en-Y gastric bypass).
* Have a BMI less than 17 kg/m^2 or more than 40 kg/m^2 at the time of screening.
* Diagnosed with a major psychiatric disorder according to the MINI.
* Have a past or current diagnosis of schizophrenia or bipolar disorder.
* At risk of suicide (C-SSRS score of 4 or higher) or have attempted suicide in the past 2 weeks.
* Have active and progressive physical illnesses (e.g., congestive heart failure, chronic obstructive pulmonary disease, acute pain), neurological disorders (e.g., cerebrovascular disease), neurodegenerative diseases (e.g., dementia, multiple sclerosis), unstable medical conditions, or a life expectancy of less than 6 months.
* Pregnant or planning to become pregnant during the trial period.
* Participated in another clinical trial within 4 weeks prior to screening.
* Have a history of alcohol or substance abuse.
* Considered by the investigator to be unsuitable for participation in this clinical trial for any other reason.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Binge Eating Frequency | from baseline (pre-use) to the 8-week point.
  Change of Binge Eating Frequency (item 14 of the Eating Disorder Examination Questionnaire, EDE-Q)

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | 8 weeks
  28 items divided into four subscales: dietary restraint, concern with eating, concern with body shape, and concern with weight. Excluding frequency questions, it assesses symptoms over the past 4 weeks on a 7-point scale from 0 to 6, where higher scores indicate more problematic eating behaviors and attitudes.
Clinical Impairment Assessment (CIA) | 8 weeks
  Purpose: Evaluates the secondary impairment in three main areas (personal, social, and cognitive) related to eating disorders.
  Format: A brief self-report tool consisting of 16 items, scored on a 4-point scale from 0 (no impairment) to 3 (high impairment).
  Interpretation: Total score ranges from 0 to 48, higher scores indicate greater personal, social, and cognitive impairment due to eating disorders.
Patient health questionnaire-9 (PHQ-9) | 8 weeks
  Purpose: Assesses symptoms of depression based on the diagnostic criteria for major depressive disorder in DSM-IV, focusing on the past two weeks.
  Format: Comprises 9 questions related to mood, sleep changes, fatigue, appetite change, guilt, worthlessness, concentration difficulty, restlessness, and suicidal thoughts, scored from 0 (not at all) to 3 (nearly every day).
  Interpretation: Higher scores indicate more severe symptoms of depression.
Generalized anxiety disorder 7-item scale (GAD-7) | 8 weeks
  Purpose: A screening tool developed to identify symptoms of generalized anxiety disorder, evaluating the severity of related anxiety or worry.
  Format: Contains 7 items, with responses ranging from 0 (not at all) to 3 (nearly every day).
  Interpretation: Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms and greater functional impairment.
The EuroQol Visual Analogue Scale (EQ-VAS) | 8 weeks
  Purpose: Measures the participant's overall health status as part of a quality of life questionnaire.
  Format: A visual analogue scale from 0 to 100. Interpretation: Higher scores represent better overall health status.
Clinical Global Impression of Improvement (CGI-I) | 8 weeks
  Purpose: Assesses the degree of improvement or worsening in a participant's overall health status at 4 weeks (Visit 3) and 8 weeks (Visit 5).
  Format: Rated on a 7-point scale, with lower scores indicating greater improvement.
  Interpretation: Designed to provide a description of change over time, emphasizing the clinician's perspective on patient progress.
Clinical Global Impression of Severity (CGI-S) | 8 weeks
  Purpose: Evaluates the overall severity of the participant's condition at baseline, 4 weeks (Visit 3), and 8 weeks (Visit 5).
  Format: A 7-point scale is used, with higher scores indicating greater disease severity.
  Interpretation: Aims to quantify the severity of the condition from a clinical standpoint, offering insight into the disorder's impact on the patient's life.

OTHER OUTCOMES:
Adherence (Compliance) to WELT-ED (applicable only to WELT-ED Group) | 8weeks
  Adherence at the 8-week mark (Visit 5) is evaluated based on the completion rate of self-monitoring food diaries and the number of logins to the app (applicable only to the experimental group).
BMI (Body Mass Index) | 8weeks
  The change in BMI from baseline (pre-use) to after 8 weeks of using the medical device (Visit 5) is assessed. BMI = weight (kg) / height (m)^2.
WELT-ED App Usage Satisfaction (applicable only to WELT-ED Group) | 8 weeks
  App usage satisfaction is assessed through a questionnaire at the 8-week mark (Visit 5) (applicable only to the experimental group).
App-Based Lifestyle and Eating Data (applicable only to WELT-ED Group) | 8weeks
  The participants' lifestyle habits (Activity data is evaluated as change of number of steps) and eating data are evaluated through self-monitoring food diaries collected via the app.
Change in Regular Meal Frequency (applicable only to WELT-ED Group) | 8 weeks
  Changes in the frequency of meals are assessed through self-monitoring food diaries collected via the app

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No